CLINICAL TRIAL: NCT05298397
Title: Pilot Study Examining Adaptation of EAT-PTSD (the MOW Protocol) for Anxious Youth
Brief Title: Pilot Study Adapting EAT-PTSD for Anxious Youth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI stopped study due to staff turnover, recruitment/scheduling problems, policy changes, will redesign
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Prudence Fisher, Research Scientist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8260
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Disorder of Childhood or Adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention - EAT (Experimental): This study has one arm (it is an open trial). All participants will receive the intervention (EAT-PTSD adapted for youth).
  Interventions: Other: EAT-PTSD adapted for youth for anxiety

INTERVENTIONS:
Other: EAT-PTSD adapted for youth for anxiety — This is an eight session (90 minute sessions) weekly experiential group treatment. The first session includes psychoeducation, orientation to treatment, a barn tour, and ends with meeting the horses. Subsequent sessions involve increasingly complex encounters and interactions with horses accompanied by feedback and direction from the treatment. Early phase treatment exercises acquaint patients with the horse, with grooming exercises, leading with a rope or a wand, and directing the horse. The middle phase furthers patients' mastery and comfort with the horse in individual and teamwork exercises. The final session includes a graduation ceremony. All intervention sessions begin with "Opening Circle" and end with "Closing Circle." Opening Circle incorporates a "grounding exercise" and is orients participants to the session to check in regarding thoughts and feelings. Closing Circle reviews lessons learned during the session, eliciting participant feedback and facilitating discussion.

SUMMARY:
The purpose of this research protocol is to adapt the Equine Assisted Therapy (EAT) protocol, which the investigators had developed to help treat PTSD (EAT-PTSD; the Man O' War (MOW) protocol), for use with adolescents who have an anxiety disorder.

The MOW protocol is an eight session, group therapy EAT protocol, which the investigators developed, piloted, revised, and tested. EAT is an alternative treatment practiced across the United States and around the world for mental health disorders, in which the horse(s) play an essential role in an experientially oriented therapeutic approach. The MOW protocol is for group EAT, with groups led by a licensed mental health provider and an "equine specialist," working with two horses and assisted by a wrangler (horse handler) to assure safety. In the open trial, the MOW protocol showed promising results in reducing the level of PTSD and Depressive symptoms in veterans with moderate to severe PTSD, was found to be safe (no adverse events), and well accepted (very few dropouts (Fisher et al., 2021)) and found evidence of neural changes (Zhu et al, 2021). As part of the MOW project, the investigators prepared a well specified treatment manual (Fisher et al, 2021) - the first of its kind in the field of EAT - and have trained others in its use.

DETAILED DESCRIPTION:
In this pilot study the investigators will explore the use/adaptation of the EAT-PTSD protocol that the investigators developed to treat veterans with Posttraumatic Stress Disorder so that it might be used with adolescents with anxiety disorders.

Potential participant Identification:

The first group of potential participants will be identified from the "waiting list" at CUCARD Westchester. Currently CUCARD clinic has very limited clinician availability and maintains a waitlist of up to 30 adolescents who are (or whose family are on their behalf) seeking treatment at CUCARD. The clinic's intake coordinator undertakes a basic screen with families who call and gets a basic description of the youth's symptoms (chief complaint), his/her address, current school, history of suicidal behavior and self-harm, violence, aggression, substance use, treatment history, previous diagnoses, medical problems, etc.

Clinic staff will review the waiting list for youth who are judged to be likely eligible, to help recruit the first group of six adolescents, with efforts made to have at least two of each gender in every group (and ideally balance groups by gender). To do this the investigators will start by preferentially selecting youth who: 1) live in closer proximity to the equestrian center which is in Brewster (using their address) and 2) do not attend the same school as other participants who have been included (i.e., one per school if possible), until the investigators fill a group.

For each potential participant, a clinic staff member will call their parents to let them know that the youth may be eligible for a new small study of the use of Equine Assisted Therapy for Youth who are anxious, that is being carried out on Wednesday afternoons (for Group 1 - for Group 2, it may be a different day), in collaboration with the Division of Child Psychiatry at Columbia. (NOTE: It is a usual practice at the clinic to "check-in" with families on the waiting list, to see how they are managing, whether they need a referral, etc.).

In the call, the staff member will 1.) stress that this is a new research study and that being in the study does not in any way affect their child's place on the waiting list, that they are being told about the study because it is something they might be interested in, and basically explain that it is group treatment, 8 sessions, that is being done at a private equestrian facility in Brewster. Parents will be asked if the clinic might give the research team their number so that they can tell them more about the study; they will also be given the number of the research team to contact if they are interested. The research team has prepared a script for the staff member to use.

For potentially eligible youth whose parents cannot be reached via phone call, a letter from CUCARD may be sent to parent/families stating the same information.

Families who approach the clinic in the next several months, will also be informed about the study, while the study is still recruiting.

The research team will also send flyers to local providers informing them about the study so that they might refer potential participants. The same procedures for eligibility described below will be used for these non CUCARD affiliated potential participants.

NOTE: if necessary, the investigators will accept adolescents currently in treatment, although the preference is that they not be in concurrent treatment.

Potential Eligibility assessment (Screening):

For those who are interested, Dr. Fisher will conduct a phone screen (20-30 minutes) with the parent to assess their child's potential eligibility) and further explaining what the protocol entails (location of barn, timing of sessions, need for reliable transport, etc.). If deemed potentially eligible, parent and youth will be invited to come to CUCARD Westchester for an assessment visit.

Clinical assessment of Eligibility Consent/assent will be obtained at the assessment visit (ideally, in person) or using the REDCap system (via zoom) by either Dr. Fisher or Dr. Crimarco (see below). The assessment visit will take 3 hours (or could be broken into two, 90-minute visits, given family preference). The clinician will do the assessment that is currently done at CUCARD Westchester for new intakes to that clinic (which includes the ADIS-C, the SCARED, PHQ Etc.) plus the GCI (focused on Anxiety), the Pediatric Anxiety Rating Scale, and the CGAS (for the latter, ratings will be made by the clinician taking all information obtained from both informants into account). (Note: clinicians evaluating the youth are "independent" - not part of the treatment team). Parent and Youth will each complete self-report measures (See outcome measures below). Findings will be discussed with the research team who will decide whether the youth should participate in the group. A report from the assessment will be given to the family.

Treatment Protocol:

As soon as four to six (ideally six) adolescents have been recruited, group treatment sessions will begin, once per week, on a weekday afternoon at Pegasus Therapeutic Riding Center in Brewster New York, until 8 sessions have been completed - given holidays, weather, etc., completing eight sessions might take longer than 8 weeks.

The treatment protocol will be based on the manualized protocol developed and tested in the MOW Project. This protocol uses a team approach with a licensed mental health professional working with an experience "equine specialist" (each with specific roles), assisted by a wrangler (horse handler) to assure safety, with two or three horses. Of note, this is protocol does not include riding the horse; all work is on the ground and the entirety of all but the first of the eight sessions take place in a round pen (large paddock). Unlike many EAT programs, the horses are rarely "at liberty," - instead they have halters and lead ropes at all time for the first four sessions, and most of the time in sessions 5-8; at no time is an individual alone with a horse who is loose. The first session includes a psychoeducation piece, first session orients patients to the treatment (rationale, description, possible benefits), provides psychoeducation (which will be altered to address youth anxiety, rather than PTSD), includes a barn tour, and ends with meeting the horses in the round-pen.

Subsequent sessions review the previous session content and introduce increasingly complex encounters and interactions with horses, with team feedback and direction. Early phase treatment exercises (sessions 2-3) acquaint patients with the horse, with grooming exercises, leading with a rope or a wand, and directing the horse. The middle phase (sessions 4-7) furthers patients' mastery and comfort with the horse in individual and teamwork exercises. For example, in the "send away" activity, patients learn to use a wand to distance the horse creating personal space. The "Join up" exercise combines previously learned individual and group activities, helping participants to demonstrate partnership with the horse and direct it mid-movement. The "tarp" exercise, in which participants must work together to maneuver one of the horses onto a tarpaulin, fosters teamwork and cooperation. The final session includes a graduation ceremony celebrating treatment progress and accomplishments. Each session ends with an opportunity for participants to review and discuss their experiences ("closing circle").

PLEASE NOTE: All sessions will be observed by Prudence Fisher, PhD. and/or Nicholas Crimarco, PhD. (If both are not at the session, the session content will be reviewed with the missing person prior to the start of the next session). Dr. Crimarco, who is a co-Investigator on this protocol, is a senior clinical staff member at CUCARD Westchester. At the end of the session, the treatment team (MHP and ES, will meet with the research team (Drs. Fisher and Crimarco) to review the session and plan for the subsequent session.

Ongoing Assessments (Baseline - See above), Midpoint, End point. At midpoint (after session 4) and after the last session, all participants will be reassessed at the CUCARD Westchester by Independent Evaluators (not part of the treatment team). These assessments will include both parent and youth reports (see assessments). The staff who undertake these assessments will have been (or will be) trained on all the assessment measures, in line with the clinic protocols in place at CUCARD, with additional training by Drs. Fisher or Crimarco on the Pediatric Anxiety Scale and CGI. These staff will not be part of the treatment team.

PLEASE NOTE: Prior to Session 1 and after Sessions 4 and 8, the research team will provide clinical information from the assessment sessions to the treatment team.

After the final sessions, Dr. Fisher and/or Dr. Crimarco will meet with each family to get feedback on what they liked or didn't like about the treatment protocol.

Criteria for Early Discontinuation:

Participants may be removed from the Protocol for any of the following reasons:

1. Requests to withdraw from the study
2. Worsening of Anxiety Symptoms at midpoint assessment as measure by the CGI at the level of 5 or greater or the PARS Global ratings. (This will be reviewed with Dr. Crimarco and/or Dr. Pulifico)
3. Clear cut deterioration in functioning as assessed by Drs. Crimarco, Pulifico, or CUCARD assessor
4. New or intercurrent illness that prevents the participant from complying with the protocol
5. Non attendance at treatment sessions. As sessions build upon one another, if a participant misses two or more sessions in row (up through session six) it is difficult to incorporate him/her back into the group.
6. Significant suicide ideation or a suicide attempt (as assessed by Drs. Crimarco, Pulifico, or CUCARD assessor)
7. Physical aggression to group members and or the horses. Upon termination from the study, participants will be provided with immediate assistance as appropriate, following CUCARD protocols, which could include referral to a different agency, hospital, etc.

Confidentiality All data collected will be kept confidential and used for research purposes only.

Patient charts will be kept in locked file cabinets identified by number rather than by name and access to research records is restricted to research staff and Federal, State, and Institutional regulatory authorities. Electronic data will be protected by password access. No names of subjects will be recorded or written on any research instrument. No participant's identifying data will be published.

The study was closed after four participants had signed consent and undergone baseline assessments, but BEFORE any had been given the intervention. This is because we were unable to find a time that worked for all four -- this is group intervention.. Thus, there are no outcome measures or results to report; the dates regarding "completion" refer to when the initial (baseline) data were collected for the fourth participant.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 13-17
* Youth lives with parent
* English speaking (youth and parent) who reside in Westchester, Putnam, Rockland, Bronx, or Manhattan Counties (in New York) OR in Connecticut
* Youth does not have a current substance use problem
* Youth is available for an "after school" group at time the EAT sessions are scheduled
* Parent understands that participation does not affect place on clinic waiting list
* Parent will be able to provide/assure transportation to equestrian center, etc.
* Current diagnosis of Social Anxiety Disorder, Separation Anxiety Disorder, Generalized Anxiety Disorder, or Unspecified Anxiety Disorder
* Parent understands the protocol, agrees to their responsibilities (providing transport, scheduling sessions), and is able to give consent
* Youth understands the protocol and consents (if age 18) or assents (if younger than age 18) of their own free will

Exclusion Criteria:

* Elevated depression, PTSD, or OCD symptoms of clinical concern
* Elevated risk for suicide/suicidal behavior based on history and current mental state
* Extreme fear of horses
* Orthopedic or other physical limitation that would prevent youth from walking unassessed and/or walking freely in ring
* Acute, unstable, or severe medical disorder (that might prohibit completing the 8 session protocol)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale - Global Ratings (PARS) | 5 minutes
  A clinician-rated measure of symptom severity and associated impairment that targets generalized anxiety disorder, social phobia, and separation anxiety disorder
Children's Global Assessment Scale (CGAS) | 2 minutes
  A clinician rating of a child's social and psychological functioning
Screen for Child Anxiety Related Disorders (SCARED) - Youth | 4 minutes
  A child self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder and social phobia
Screen for Child Anxiety Related Disorders (SCARED) - Parent | 4 minutes
  A parent/other administered scale that aids in the diagnosis of panic disorder/significant somatic symptoms, generalized anxiety disorder, separation anxiety disorder, social anxiety disorder, and significant school avoidance
Clinical Global Impressions - Improvement Scale (CGI-I) | 2 minutes
  A scale that rates the degree of clinical improvement at the time of assessment, relative to how the patient was at entry (Score from 1-7)

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule - Child and Parent (ADIS-C) | 160 minutes
  A semistructured interview used to assess for Diagnostic and Statistical Manual of Mental Disorders anxiety disorder diagnoses on the basis of both child and parent report
Columbia Impairment Scale - Parent Form | 2 minutes
  A measure of general impairment in various functional domains, including relations with family members at home, relations with peers, academic or occupational functioning, and involvement in general interests and activities
Mood and Feelings Questionnaire - Parent Long Form | 5 minutes
  A series of 33 descriptive phrases regarding how the subject has been feeling or acting recently, used to screen for depression in children and young people aged 6 to 19
Mood and Feelings Questionnaire - Youth Long Form | 5 minutes
  A series of 33 descriptive phrases regarding how the subject has been feeling or acting recently, used to screen for depression in children and young people aged 6 to 19
Patient-Reported Outcomes Measurement Information System (PROMIS): Short Form 8A - Family Relationships (Parent) | 2 minutes
  A scale to measure patient reported outcomes for clinical research and practice - completed by parent
Patient-Reported Outcomes Measurement Information System (PROMIS): Short Form 8A - Family Relationships (Child) | 2 minutes
  A scale to measure patient reported outcomes for clinical research and practice - completed by youth
Adolescent Self Esteem Questionnaire | 3 minutes
  A 13-item measure of global self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Prudence Fisher, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - 1051 Riverside Drive, New York, New York
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu X, Suarez-Jimenez B, Zilcha-Mano S, Lazarov A, Arnon S, Lowell AL, Bergman M, Ryba M, Hamilton AJ, Hamilton JF, Turner JB, Markowitz JC, Fisher PW, Neria Y. Neural changes following equine-assisted therapy for posttraumatic stress disorder: A longitudinal multimodal imaging study. Hum Brain Mapp. 2021 Apr 15;42(6):1930-1939. doi: 10.1002/hbm.25360. Epub 2021 Feb 5. PMID 33547694
- [Background] Fisher PW, Lazarov A, Lowell A, Arnon S, Turner JB, Bergman M, Ryba M, Such S, Marohasy C, Zhu X, Suarez-Jimenez B, Markowitz JC, Neria Y. Equine-Assisted Therapy for Posttraumatic Stress Disorder Among Military Veterans: An Open Trial. J Clin Psychiatry. 2021 Aug 31;82(5):21m14005. doi: 10.4088/JCP.21m14005. PMID 34464523
- [Background] Arnon S, Fisher PW, Pickover A, Lowell A, Turner JB, Hilburn A, Jacob-McVey J, Malajian BE, Farber DG, Hamilton JF, Hamilton A, Markowitz JC, Neria Y. Equine-Assisted Therapy for Veterans with PTSD: Manual Development and Preliminary Findings. Mil Med. 2020 Jun 8;185(5-6):e557-e564. doi: 10.1093/milmed/usz444. PMID 32034416